CLINICAL TRIAL: NCT07363954
Title: A Clinical Study on the Safety, Efficacy, and Pharmacokinetics of STR-P004 for the Treatment of Immune-Mediated Kidney Diseases
Brief Title: To Evaluate the Safety and Tolerability of STR-P004 for the Treatment of Immune-mediated Kidney Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Starna Therapeutics (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STR-P004-005
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose1 (Experimental)
  Interventions: Drug: STR-P004 dose group

INTERVENTIONS:
Drug: STR-P004 dose group — Three dose groups are planned: DL1 XXmg/kg, DL2 XXmg/kg, DL3 XX mg/kg. Starting dose is XX mg/kg.

SUMMARY:
This is a single-center, non-randomized, open-label, single-arm exploratory clinical study, using Bayesian Optimal Interval (BOIN) design. Three dose groups are planned: DL1 XX mg/kg, DL2 XXmg/kg, DL3 XXmg/kg. Starting dose is XX mg/kg. Each treatment cycle is 28 days, with 4 infusions on D1, D4, D7, D10; 1-2 cycles. The investigator may escalate to higher doses to further explore safety and efficacy of STR-P004 based on preliminary safety data, efficacy information, and PK/PD parameters obtained.

DETAILED DESCRIPTION:
This is a single-center, non-randomized, open-label, single-arm exploratory clinical study, using Bayesian Optimal Interval (BOIN) design. Three dose groups are planned: DL1 XXmg/kg, DL2 XXmg/kg, DL3 XX mg/kg. Starting dose is XX mg/kg. Each treatment cycle is 28 days, with 4 infusions on D1, D4, D7, D10; 1-2 cycles. The investigator may escalate to higher doses to further explore safety and efficacy of STR-P004 based on preliminary safety data, efficacy information, and PK/PD parameters obtained.

After dose escalation is completed, the investigator and collaborator may select 1 or 2 dose groups for an expansion cohort study (or during dose escalation). Each dose group will enroll an additional 3-6 subjects to evaluate efficacy and determine the RP2D.

This study aims to determine the safety, tolerability, and RP2D of STR-P004 in subjects with immune-mediated kidney diseases. The study will also evaluate the PK characteristics of STR-P004 and provide preliminary efficacy observations

ELIGIBILITY:
Inclusion Criteria:

* 1. Willing and able to provide written informed consent. 2. Age between 18 and 75 years (inclusive). 3. Confirmed CD19-positive B cell expression in peripheral blood by flow cytometry.

  4.Adequate organ function:
  1. Bone marrow function: defined as absolute neutrophil count (ANC) ≥1500 /μL, absolute lymphocyte count (ALC) ≥100 /μL, hemoglobin (Hb) ≥80 g/L, platelet count (PLT) ≥50,000 /μL. Use of transfusions or growth factors to meet these requirements within 7 days prior to screening is not allowed.
  2. Liver function: defined as alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN, total bilirubin <1.5×ULN (<3.0×ULN for subjects with Gilbert's syndrome).
  3. Coagulation function: defined as International Normalized Ratio (INR) or activated partial thromboplastin time (APTT) ≤1.5×ULN.
  4. Pulmonary function: defined as ≤ CTCAE Grade 1 dyspnea and oxygen saturation (SpO2) ≥92% on room air at rest (by pulse oximetry).

     5. Women of childbearing potential (defined as all women physiologically capable of becoming pregnant) must agree to use highly effective contraceptive methods from signing ICF until 1 year after STR-P004 infusion (including during study treatment interruption). Male subjects with partners of childbearing potential must agree to use effective barrier contraception methods for 1 year after STR-P004 infusion and should not donate semen or sperm during the entire study period.

     6. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) test at screening and within 48 hours prior to STR-P004 infusion. Women who have undergone sterilization or are postmenopausal for at least 2 years are considered not of childbearing potential.

     Exclusion Criteria:
* 1. Any clinically significant underlying disease, other than SLE/LN, AAV/AAGN, Anti-GBM Disease, MN, APSN, and IgG4-RKD, that, in the investigator's opinion, poses a safety risk or problem.

  2. Rapidly progressive glomerulonephritis not related to SLE/LN, AAV/AAGN, Anti-GBM Disease, MN, APSN, and IgG4-RKD, defined as ≥50% reduction in eGFR within 3 months since diagnosis.

  3. Other uncontrolled serious conditions not directly related to the disease prior to screening, such as severe hemolytic anemia, severe thrombocytopenic purpura, severe agranulocytosis, severe myocardial damage, severe pneumonia or pulmonary hemorrhage, severe hepatitis, severe vasculitis, active central nervous system symptoms including cerebrovascular accident, aneurysm, epilepsy, convulsions/seizures, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT, SAE, and Treatment-Emergent Adverse Events (TEAE). | 3 months